CLINICAL TRIAL: NCT05092152
Title: Propofol Versus Ketamine for Rapid Sequence Intubation in Critically Ill Patients: A Randomized, Multicenter, Unblinded, Clinical Trial
Brief Title: Propofol Versus Ketamine for Rapid Sequence Intubation in Critically Ill Patients
Acronym: PROMINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Flavia Ribeiro Machado, Chair of Critical Care Department, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMINE
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Acute Respiratory Failure
Keywords: rapid sequence intubation; intubation; airway management; propofol; ketamine; hypnotics
MeSH Terms: interventions — Esketamine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Active Comparator)
  Interventions: Drug: Propofol
- Ketamine (Experimental)
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — 2 mg per kilogram of body weight
  Arms: Ketamine
Drug: Propofol — 1.5 mg per kilogram of body weight
  Arms: Propofol

SUMMARY:
Rapid-sequence intubation is routinely performed in critically ill patients. It is unclear whether different sedative agents may influence short-term outcomes after intubation, specially hemodynamic stability.

DETAILED DESCRIPTION:
The optimal and safest hypnotic agent for rapid sequence intubation in critically ill patients remains uncertain. Factors such as hypovolemia, vasoplegia, hypoxemia, and acidosis can influence the efficacy and safety of induction agents. Propofol is commonly used for this purpose; however, it is associated with the risk of exacerbating hypotension. Ketamine, which has a more favorable hemodynamic profile, may offer a safer alternative in these patients. Objective: To assess whether ketamine is a safer alternative to propofol for rapid sequence intubation by reducing the incidence of hypotension during induction in critically ill patients.

Methods: This will be a randomized, open-label, pragmatic, bicenter study. A total of 170 critically ill patients requiring endotracheal intubation in the intensive care unit will be randomly assigned to receive either ketamine or propofol as the hypnotic agent. Randomization will be conducted using RedCap with a 1:1 ratio and variable block sizes, stratified by study site and vasopressor use during intubation. Results: The primary outcome will be the occurrence of hypotension, defined as the lowest mean arterial pressure recorded within the first 10 minutes following induction. Secondary outcomes, assessed within 1 hour post-induction, include mortality, incidence of cardiopulmonary arrest, the occurrence of severe hypotension (systolic blood pressure <80mmHg), the occurrence of severe hypoxemia (oxygen saturation < 85%), and the number of intubation attempts. Conclusion: The PROMINE study will provide valuable evidence to guide the selection of hypnotic agents for rapid sequence intubation in critically ill patients. It will contribute to a better understanding of the hemodynamic effects associated with propofol and ketamine in this context, potentially informing clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old
* Physician indicated intubation

Exclusion Criteria:

* Pregnancy
* Intubation during cardiac arrest
* Known of suspected intracranial hypertension
* Know allergy to any of the study drugs (lidocaine, fentanyl, propofol, ketamine, or rocuronium)
* Bradycardia (heart rate below 50 beats per minute) or atrioventricular block without a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2021-10-23 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Lowest mean blood pressure | Ten minutes after induction
  Lowest mean blood pressure

SECONDARY OUTCOMES:
Average MAP within the first hour after induction | 1 hour
  Average MAP within the first hour after induction
Early death | 01 hour
  Death within one hour of intubation
Cardiac arrest | 01 hour
  Cardiac arrest requiring resuscitation
Severe hypotension | 01 hour
  Systolic blood pressure below 80 mmHg
Severe hypoxemia | 01 hour
  Peripheral oxygen saturation below 85%
Time for successful intubation | 01 hour
  Time for successful intubation

OTHER OUTCOMES:
The number of intubation attempts | 01 hour
  The number of intubation attempts
The highest heart rate (HR) within one hour after induction | 01 hour
  The highest heart rate (HR) within one hour after induction
The total dose of vasopressors administered within the first 24 hours, using noradrenaline equivalent dose | 24 hours after intubation
  Cumulative, in milligrams, dose of vasopressors used
Mean change in vasopressor dose (norepinephrine equivalent) from baseline to hour 1 | 01 hour
  Mean change in vasopressor dose (norepinephrine equivalent) from baseline to hour 1
Ventilator-free days within the first 7 days | 07 days
  Ventilator-free days within the first 7 days, defined as the number of days on which individuals are able to breathe spontaneously without any invasive ventilatory assistance, ascribing zero days to those who die, within 7 days.
Mortality at day 7 | Seven days
  Mortality at day 7
ICU mortality | 60 days
  Mortality in the Intensive Care Unit
Hospital mortality | 60 days
  Mortality in hospital
Number of participants with Hypertension, defined as SBP > 180 mmHg | the first 10 minutes
  Number of participants with Hypertension, defined as SBP > 180 mmHg Safety outcomes during the first 10 minutes
Number of participants with laryngospasm, as reported by the physician in charge of intubation | 10 minutes
  Laryngospasm, as reported by the physician in charge of intubation - safety outcome
Number of participants with bradycardia, defined as HR < 45 bpm | 10 minutes
  Bradycardia, defined as HR < 45 bpm - safety outcome
Number of participants with arrhythmias | 10 minutes
  Arrhythmias - safety outcome
Number of participants with bronchoaspiration | 10 minutes
  Bronchoaspiration, defined as the presence of gastric content aspirated into the airway during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Flavia R Machado, MD, PhD, Study Chair — Federal University of São Paulo; Raysa Schmidt, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be share after publication upon resonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication
Access Criteria: Upon reasonable request

REFERENCES:
- [Derived] Schmidt RC, Zampieri FG, Ramos FJDS, Serra FSC, Damiani LP, Freitas FGR, Machado FR. Prospective, randomized, controlled trial comparing PROpofol versus KetaMINE in rapid sequence intubation in critically ill patients (PROMINE): protocol paper and statistical analysis plan. Crit Care Sci. 2025 Nov 17;37:e20250133. doi: 10.62675/2965-2774.20250133. eCollection 2025. PMID 41259542